CLINICAL TRIAL: NCT06831760
Title: A Randomized, Controlled Clinical Trial Evaluating the Efficacy of Type-I Collagen-based Skin Substitute vs. Dehydrated Human Amnion/Chorion Membrane in the Treatment of Venous Leg Ulcers
Brief Title: A RCT Evaluating Efficacy of Type-I Collagen Skin Substitute vs. Human Amnion Membrane in Treatment of Venous Leg Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Naveen Narayan MS, MCh (Plastic Surgery) (Other)
Responsible Party: Sponsor-Investigator, Dr Naveen Narayan MS, MCh (Plastic Surgery), Professor & HoD, Department of Plastic Reconstructive & Aesthetic Surgery, Adichunchanagiri Institute of Medical Sciences, B G Nagara
Organization: Adichunchanagiri Institute of Medical Sciences, B G Nagara (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIMS/IEC/004/2025
Record Dates: First submitted 2025-01-27; First posted 2025-02-18 (Actual); Results first posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Venous Leg Ulcers
Keywords: venous leg ulcer; chronic leg ulcer; leg ulcer; skin substitute; high purity type-I collagen; dehydrated human amnion / chorion membrane
MeSH Terms: conditions — Varicose Ulcer; Leg Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SOC and Type-I Collagen-based Skin Substitute (Other): The SOC in this study is wound care covering with High Purity Type-I Collagen-based Skin Substitute applied weekly or as needed followed by a padded 3-layer dressing
  Interventions: Device: SOC and Type-I Collagen-based Skin Substitute
- SOC and Human Amnion/Chorion Membrane (Other): The SOC in this study is wound care covering with Dehydrated Human Amnion/Chorion Membrane followed by a padded 3-layer dressing
  Interventions: Device: SOC and Human Amnion/Chorion Membrane

INTERVENTIONS:
Device: SOC and Type-I Collagen-based Skin Substitute — The SOC in this study is wound care covering with High Purity Type-I Collagen-based Skin Substitute applied weekly or as needed followed by a padded 3-layer dressing comprised of first layer - non-adherent and porous, second layer - absorbent 4x4 gauze pads & third layer - soft roll and compressive wrap
  Arms: SOC and Type-I Collagen-based Skin Substitute
Device: SOC and Human Amnion/Chorion Membrane — The SOC in this study is wound care covering with Dehydrated Human Amnion/Chorion Membrane followed by a padded 3-layer dressing comprised of first layer - non-adherent and porous, second layer - absorbent 4x4 gauze pads & third layer - soft roll and compressive wrap
  Arms: SOC and Human Amnion/Chorion Membrane

SUMMARY:
Venous leg ulcers are chronic wounds caused by venous insufficiency, leading to significant morbidity. The purpose of this randomized, controlled study is to evaluate the safety and efficacy of the application of Type-I Collagen-based Skin Substitute (HPTC) vs. Dehydrated Human Amnion/Chorion Membrane (dHCAM) in the treatment of VLUs and to compare their efficacy.

DETAILED DESCRIPTION:
Venous leg ulcers (VLUs) are chronic wounds caused by venous insufficiency, leading to significant morbidity. Current treatment options often include compression therapy, wound debridement, and advanced dressings. Despite advances in wound care, effective treatment remains challenging. The purpose of this randomized, controlled study is to evaluate the safety and efficacy of the application of Type-I Collagen-based Skin Substitute (HPTC) vs. Dehydrated Human Amnion/Chorion Membrane (dHCAM) in the treatment of VLUs and to compare the efficacy of these two advanced wound care modalities in accelerating VLU healing.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be at least 18 years of age or older.
2. Subjects must have a diagnosis of a venous leg ulcer (confirmed by clinical and duplex ultrasound evaluation).
3. At enrolment subjects must have a target VLU with a minimum surface area of 2.0 cm2 and a maximum surface area of 25.0 cm2 measured post debridement using a ruler to measure wound area.
4. The target ulcer must have been present for a minimum of 4 weeks and a maximum of 52 weeks of standard of care prior to the initial screening visit.
5. The target ulcer must be located on the foot, ankle and lower leg region.
6. The target ulcer must be full thickness on the foot or ankle that does not probe to bone.
7. Adequate circulation to the affected foot as documented by any of the following methods performed within 3 months of the first screening visit:

i. TCOM ≥30 mmHg ii. ABI between 0.7 and 1.3 iii. PVR: Biphasic iv. TBI ˃0.6 v. As an alternative arterial, Doppler ultrasound can be performed evaluating for biphasic dorsalis pedis and posterior tibial vessels at the level of the ankle of the target extremity.

h. If the subject has two or more ulcers, they must be separated by at least 2 cm. The largest ulcer satisfying the inclusion and exclusion criteria will be designated as the target ulcer.

i. The subject must consent to using the prescribed off-loading method for the duration of the study.

j. The subject must agree to attend the twice-weekly/weekly study visits required by the protocol.

k. The subject must be willing and able to participate in the informed consent process.

l. Patients must have read and signed the IRB approved ICF before screening procedures are undertaken.

Exclusion Criteria:

1. A subject known to have a life expectancy of <6 months
2. If the target ulcer is infected or if there is cellulitis in the surrounding skin.
3. Presence of osteomyelitis or exposed bone, probes to bone or joint capsule on investigator's exam or radiographic evidence.
4. A subject that has an infection in the target ulcer that requires systemic antibiotic therapy.
5. A subject receiving immunosuppressants (including systemic corticosteroids at doses greater than 10 mg of Prednisone per day or equivalent) or cytotoxic chemotherapy.
6. Topical application of steroids to the ulcer surface within one month of initial screening.
7. A subject with a previous partial amputation on the affected foot is excluded if the resulting deformity impedes proper offloading of the target ulcer.
8. A subject with autoimmune or connective tissue disorders.
9. A subject with malignant wounds or non-venous ulcers.
10. A subject with a serum creatinine ≥ 3.0mg/dL within 6 months of the initial screening visit.
11. Women who are pregnant or considering becoming pregnant within the next 6 months and those who are breast feeding.
12. A subject with end stage renal disease requiring dialysis.
13. A subject who participated in a clinical trial involving treatment with an investigational product within the previous 30 days.
14. A subject who, in the opinion of the Investigator, has a medical or psychological condition that may interfere with study assessments.
15. A subject treated with hyperbaric oxygen therapy or a Cellular and/or Tissue Product (CTP) in the 30 days prior to the initial screening visit.
16. History of autoimmune disease, malignancy, or uncontrolled diabetes (HbA1c >10%).
17. Allergy to components of High Purity Type-I Collagen-based Skin Substitute or Dehydrated Human Amnion/Chorion Membrane.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prema Dhanraj, MS, MCh, Study Chair — Rajarajeshwari Medical College and Hospital
Locations (1):
- Adichunchanagiri Institute of Medical Sciences, Mandya, Karnataka, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bianchi C, Cazzell S, Vayser D, Reyzelman AM, Dosluoglu H, Tovmassian G; EpiFix VLU Study Group. A multicentre randomised controlled trial evaluating the efficacy of dehydrated human amnion/chorion membrane (EpiFix(R) ) allograft for the treatment of venous leg ulcers. Int Wound J. 2018 Feb;15(1):114-122. doi: 10.1111/iwj.12843. Epub 2017 Oct 11. PMID 29024419
- [Background] Narayan N, Gowda S, Shivannaiah C. A Randomized Controlled Clinical Trial Comparing the Use of High Purity Type-I Collagen-Based Skin Substitute vs. Dehydrated Human Amnion/Chorion Membrane in the Treatment of Diabetic Foot Ulcers. Cureus. 2024 Dec 5;16(12):e75182. doi: 10.7759/cureus.75182. eCollection 2024 Dec. PMID 39649230
- [Background] Serena TE, Carter MJ, Le LT, Sabo MJ, DiMarco DT; EpiFix VLU Study Group. A multicenter, randomized, controlled clinical trial evaluating the use of dehydrated human amnion/chorion membrane allografts and multilayer compression therapy vs. multilayer compression therapy alone in the treatment of venous leg ulcers. Wound Repair Regen. 2014 Nov-Dec;22(6):688-93. doi: 10.1111/wrr.12227. Epub 2015 Jan 8. PMID 25224019

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 26
  Male | 20 | 14 | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  India | 30 | 30 | 60
Ulcer duration [Mean (Standard Deviation); unit: Months] | 2.13 (1.14) | 2.43 (1.28) | 2.28 (1.21)
Ulcer size [Mean (Standard Deviation); unit: square centimeters] | 14.84 (1.87) | 15.19 (1.91) | 15.02 (1.89)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Wound Area Change
Description: Percentage wound area change from week 1 through week 7 measured manually with digital photography
Time Frame: 7 Weeks
Measure: Mean (Standard Deviation); unit: percentage wound area reduction
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 30 | 30
percentage wound area reduction | 78.9 (17.8) | 65.4 (7.9)

2. Primary Outcome: Histopathological Parameters - Vascular Infiltration
Description: Histopathological Assessment - Before application and on the 5th day post-application of either HPTC or dHCAM, a 2mm punch biopsy was obtained from the wound edge extending into the wound bed under local anaesthesia. Serial sections of 4μm thickness were prepared and stained with Hematoxylin and Eosin (H&E) for general morphology.
  Vascular Infiltration: Assessed by counting new blood vessels per High Power Field (hpf) (0-3 scale) 0: Minimal vascular ingrowth (<5 vessels/hpf)
  1. Mild infiltration (5-10 vessels/hpf)
  2. Moderate infiltration (11-20 vessels/hpf)
  3. Abundant infiltration (>20 vessels/hpf)
  (0-worse; 3-better)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale (0-worse; 3-better)
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 30 | 30
score on a scale (0-worse; 3-better) | 2.73 (0.45) | 1.87 (0.68)

3. Primary Outcome: Histopathological Parameters - Neo-epithelialization
Description: Before application and on the 5th day post-application of either HPTC or dHCAM, a 2mm punch biopsy was obtained from the wound edge extending into the wound bed under local anaesthesia. Serial sections of 4μm thickness were prepared and stained with: Hematoxylin and Eosin (H&E) for general morphology.
  Neo-epithelialization: Measured as epithelial migration distance from wound edge (0-3 scale) 0: No epithelial migration
  1. Minimal migration (<25% wound coverage)
  2. Moderate migration (25-75% coverage)
  3. Extensive migration (>75% coverage)
  (0-worse; 3-better)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale (0-worse; 3-better)
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 30 | 30
score on a scale (0-worse; 3-better) | 2.67 (0.48) | 1.63 (0.72)

4. Primary Outcome: Histopathological Parameters - Fibroblast Activity
Description: Before application and on the 5th day post-application of either HPTC or dHCAM, a 2mm punch biopsy was obtained from the wound edge extending into the wound bed under local anaesthesia. Serial sections of 4μm thickness were prepared and stained with: α-SMA immunohistochemistry for fibroblast activity.
  Fibroblast Activity: Quantified by counting α-SMA positive fibroblasts per HPF and assessment of fibroblast morphology (0-3 scale) 0: Sparse, inactive fibroblasts
  1. Moderate cellularity, minimal matrix production
  2. High cellularity, active-matrix synthesis
  3. Very high activity with extensive matrix deposition
  (0-worse; 3-better)
Time Frame: 5 Days
Measure: Mean (Standard Deviation); unit: score on a scale (0-worse; 3-better)
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 30 | 30
score on a scale (0-worse; 3-better) | 2.80 (0.41) | 1.93 (0.64)

5. Primary Outcome: Histopathological Parameters - Capillary Density
Description: Histopathological Assessment - Before application and on the 5th day post-application of either HPTC or dHCAM, a 2mm punch biopsy was obtained from the wound edge extending into the wound bed under local anaesthesia.
  Serial sections of 4μm thickness were prepared and stained with: CD31 immunohistochemistry for capillary density evaluation Capillary Density: Evaluated using CD31 staining, counted as vessels per mm² of tissue
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: number of vessels per mm² of tissue
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 30 | 30
number of vessels per mm² of tissue | 47.3 (8.2) | 28.7 (9.6)

6. Primary Outcome: Histopathological Parameters - Inflammatory Response
Description: Histopathological Assessment - Before application and on the 5th day post-application of either HPTC or dHCAM, a 2mm punch biopsy was obtained from the wound edge extending into the wound bed under local anaesthesia.
  Serial sections of 4μm thickness were prepared and stained with: Hematoxylin and Eosin (H&E) for general morphology Inflammatory Response: Graded semi-quantitatively (0-3 scale) 0: Minimal inflammatory infiltrate
  1. Mild chronic inflammation
  2. Moderate mixed inflammation
  3. Severe acute inflammation
  (0-worse; 3-better)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale (0-worse; 3-better)
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 30 | 30
score on a scale (0-worse; 3-better) | 1.23 (0.43) | 2.17 (0.59)

7. Primary Outcome: Histopathological Parameters - Collagen Deposition
Description: Histopathological Assessment - Before application and on the 5th day post-application of either HPTC or dHCAM, a 2mm punch biopsy was obtained from the wound edge extending into the wound bed under local anaesthesia.
  Serial sections of 4μm thickness were prepared and stained with: Masson's Trichrome for collagen assessment Collagen Deposition: Assessed using Masson's Trichrome staining (0-3 scale) 0: Minimal collagen matrix
  1. Loose, immature collagen
  2. Moderate organized collagen
  3. Dense, mature collagen architecture
  (0-worse; 3-better)
Time Frame: 5 days
Measure: Mean (Standard Deviation); unit: score on a scale (0-worse; 3-better)
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 30 | 30
score on a scale (0-worse; 3-better) | 2.63 (0.49) | 1.77 (0.63)

8. Secondary Outcome: Time to Achieve Complete Wound Closure
Description: The time to achieve complete wound closure of the target ulcer by the end of 7 weeks
Time Frame: 7 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 30 | 30
days | 42.6 (9.8) | 46.2 (8.7)

9. Secondary Outcome: Percentage of Subjects to Obtain Complete Closure
Description: The percentage of subjects that obtain complete closure over the 7 week treatment period
Time Frame: 7 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 30 | 30
Participants | 21 | 13

10. Secondary Outcome: Number of Patients Requiring Repeated Application
Description: Number of patients requiring repeated applications of the Advanced Skin Substitute & Human Amnion/Chorion Membrane used to obtain wound closure
Time Frame: 6 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 30 | 30
Participants | 8 | 13

11. Secondary Outcome: Intervention Related Adverse Events
Description: Number of participants with intervention related adverse events related to the intervention (e.g., infection, allergic reactions)
Time Frame: 6 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 30 | 30
Participants
  No adverse event | 28 | 27
  Mild local reaction | 2 | 3
  Severe adverse events | 0 | 0

12. Other Pre Specified Outcome: Change in Pain
Description: Change in pain measured by a Visual Analog Scale with score range from 0 to 10, wherein 0="no pain" to 10="severe pain"
Time Frame: 7 weeks including 1-week follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 30 | 30
score on a scale
  Week 0 | 4.9 (1.7) | 4.6 (1.5)
  Week 1 | 2.9 (1.5) | 3.2 (1.6)
  Week 2 | 3.7 (1.3) | 3.4 (1.4)
  Week 3 | 2.8 (1.5) | 3.0 (1.3)
  Week 4 | 2.8 (1.5) | 3.2 (1.5)
  Week 5 | 2.7 (1.4) | 2.8 (1.2)
  Week 6 | 2.8 (1.6) | 3.0 (1.4)
  Week 7 | 2.9 (1.3) | 2.8 (1.5)

13. Other Pre Specified Outcome: Improvement in Quality of Life
Description: Change in quality of life assessed using the Wound-QoL questionnaire measured as 'not at all', 'a little', 'moderately', 'quite a lot' and 'very much' for 17 questions and total number of patients who reported improvement in Quality of Life was measured
Time Frame: 7 weeks including 1-week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 30 | 30
Participants | 21 | 12

14. Other Pre Specified Outcome: Healed Wound Appearance Assessment Using Manchester Scar Scale
Description: The resultant new skin is assessed and documented at each visit using the Manchester Scar Scale (MSS) assessing:
  1. Colour: Perfect - 1, Slight mismatch - 2, Obvious mismatch - 3, Gross mismatch - 4
  2. Finish: Matte - 1, Shiny - 2
  3. Contour: Flush with surrounding skin - 1, Slightly proud / indented - 2, Hypertrophic - 3, Keloid - 4
  4. Distortion: None -1, Mild - 2, Moderate - 3, Severe - 4
  Lower score denotes a better outcome using the MSS (range: 4-14). In the study, scores were categorized as such:
  1. Excellent: Scores 4 and 5
  2. Good: Scores from 6 to 8
  3. Fair: Scores from 9 to 11
  4. Poor: Scores from 12 to 14
Time Frame: 7 weeks including 1-week follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
Number analyzed (Participants) | 30 | 30
Participants
  Excellent | 2 | 0
  Good | 18 | 11
  Fair | 10 | 14
  Poor | 0 | 5

ADVERSE EVENTS:
Time Frame: 7 Weeks including 1 week follow up
Description: All the study participants were considered at risk for adverse events.
Arm/Group | SOC and Type-I Collagen-based Skin Substitute | SOC and Human Amnion/Chorion Membrane
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 2/30 | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SOC and Type-I Collagen-based Skin Substitute (N=30) | SOC and Human Amnion/Chorion Membrane (N=30)
Infections (Infections and infestations) | 0 | 0
Mild local reaction (Immune system disorders) | 2 | 3

LIMITATIONS AND CAVEATS:
Single-centre design may limit generalizability to other healthcare settings and populations.

Relatively short follow-up period (7 weeks), while sufficient for assessing acute healing outcomes, may not capture long-term outcomes, recurrence rates or durability of treatment effects. T Study was not completely blinded due to the nature of the interventions Study included a specific range of wound sizes and may not be generalizable to very large wounds.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2025-07-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT06831760/Prot_006.pdf
  • Statistical Analysis Plan (2025-07-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT06831760/SAP_007.pdf